CLINICAL TRIAL: NCT07270588
Title: MOBACT: An Internet-Based Guided Self-Help Intervention Based on Acceptance and Commitment Therapy for Chronic Pain
Brief Title: MobACT: An Internet-Based Intervention for Chronic Pain Patients
Acronym: MobACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: IRCCS Policlinico di Sant'Orsola, University Alma Mater Studiorum of Bologna, Italy (Unknown); Università degli studi di Verona (Unknown); Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gianluca Castelnuovo, Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUP J53D23008130008
Record Dates: First submitted 2025-09-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Internet-based intervention; clinical psychology; acceptance and commitment therapy
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7-weeks Internet-based interventions (Experimental): Participants allocated to the experimental group will be asked to complete one module per week, each based on the core principles of Acceptance and Commitment Therapy (ACT). The treatment program consists of seven modules delivered weekly over a total duration of seven weeks. The content of the modules will cover the following topics:
  1. Creative hopelessness
  2. Willingness and acceptance of pain
  3. Defusion from negative thoughts
  4. Committed action and values
  5. Values and goal setting
  6. Willingness exercises
  7. Maintenance of learned strategies.
  Interventions: Other: Internet-based intervention
- 7-Weeks Waiting list (No Intervention): Participants allocated to the waiting list control group will not receive the intervention during the initial seven-week study period. However, they will be granted full access to the treatment program after the seven weeks have elapsed.

INTERVENTIONS:
Other: Internet-based intervention — Participants allocated to the experimental group will be asked to complete one module per week, each based on the core principles of Acceptance and Commitment Therapy (ACT). The treatment program consists of seven modules delivered weekly over a total duration of seven weeks. The content of the modules will cover the following topics: 1. Creative hopelessness 2. Willingness and acceptance of pain 3. Defusion from negative thoughts 4. Committed action and values 5. Values and goal setting 6. Willingness exercises 7. Maintenance of learned strategies.
  Arms: 7-weeks Internet-based interventions

SUMMARY:
Chronic Pain (CP) is a condition characterized by pain that lasts or recurs for more than three months in one or more parts of the body. This type of pain is often accompanied by emotional distress and difficulties in daily functioning, which can interfere with a person's ability to carry out everyday activities and maintain social roles. As a result, it places a considerable burden not only on individuals but also on national healthcare systems, due to both direct medical costs and indirect costs such as reduced work productivity and increased use of health services.

Traditional treatments for CP, such as medications and surgical procedures, often fail to provide sufficient relief or significantly improve the quality of life of those affected. This has led to growing interest in alternative approaches that can offer more lasting and comprehensive support. In this context, psychological therapies have gained increasing attention, particularly Acceptance and Commitment Therapy, or ACT. This therapeutic approach focuses not only on the reduction of physical symptoms but also on helping people accept their pain as part of their lived experience. The goal is to promote emotional well-being and improve overall functioning by increasing what is known as psychological flexibility.

ACT is particularly relevant for people suffering from CP, as it helps them lead a meaningful life despite the presence of pain. Instead of avoiding or fighting the pain, individuals are encouraged to accept it while committing to actions that align with their personal values. This process supports emotional regulation and encourages engagement in activities that bring a sense of purpose and satisfaction. However, access to this type of psychological intervention remains limited in many contexts. Barriers such as long waiting lists, lack of trained professionals, geographic distance from treatment centers, stigma associated with psychological therapy, and patients' physical limitations often make it difficult for those in need to receive adequate care.

In response to these challenges, recent years have seen the development of new forms of digital health support. In particular, internet-delivered self-help programs have emerged as a promising solution for the treatment of CP. These programs can reach individuals who might otherwise be unable to access care and offer a flexible, low-cost, and convenient alternative to traditional face-to-face therapy. Research has shown that ACT can be effectively adapted and delivered online, allowing people to benefit from its therapeutic principles in a format that fits their needs and lifestyles.

The current study aims to evaluate the effectiveness of a guided online self-help program based on Acceptance and Commitment Therapy for individuals with CP. The program is designed to help participants accept their pain and focus on improving their quality of life through value-based actions. The study will also explore the psychological mechanisms that may explain how and why the intervention works, with the goal of improving the design and delivery of future programs. Furthermore, the study will examine the cost-effectiveness of this type of digital intervention, in order to assess its potential for broader implementation within public health systems. By increasing access to evidence-based psychological care through digital platforms, this research seeks to contribute to more effective, inclusive, and sustainable treatment options for those living with chronic pain.

DETAILED DESCRIPTION:
Introduction

Chronic Pain (CP) is pain that persists or recurs for more than three months in one or more anatomical regions, and is characterized by significant emotional distress (anxiety, anger/frustration, or depressed mood) and/or functional disability (interference with daily life activities and reduced participation in social roles), which cannot be more accurately explained by other diagnoses. Pain is defined as an unpleasant sensory and emotional experience associated with, or resembling that associated with, actual or potential tissue damage, as reported in the International Classification of Diseases (ICD-11).

Conditions such as widespread chronic pain, complex regional pain syndrome, primary chronic headache, chronic visceral pain, and chronic musculoskeletal pain affect nearly 20% of the population and represent leading causes of disability worldwide. CP is associated with reduced quality of life, decreased work productivity, and increased use of medications and healthcare services, representing a substantial economic and social burden with significant direct and indirect costs. Consequently, effective management of CP is crucial.

Chronic Pain is multifactorial: biological, psychological, and social factors all contribute to the pain syndrome. Therefore, pharmacological and surgical approaches alone are often ineffective in alleviating pain or improving physical and emotional functioning, highlighting the central importance of psychotherapy for this population.

The emotional distress of individuals with CP has been linked to pain-related coping styles. Feelings of depression, anxiety, anger, and fear are bidirectionally associated with the patient's pain experience. According to the fear-avoidance model, these factors influence pain intensity and pain-related disability, together with processes such as pain catastrophizing (i.e., a cluster of maladaptive cognitions and emotions arising in response to pain states) and pain-related fear, through avoidance behaviors. Avoidance behaviors, such as activity restriction, may lead to physical deconditioning and further reduced quality of life, producing a self-perpetuating vicious cycle.

Conversely, treatments based on Acceptance and Commitment Therapy (ACT) effectively assist patients in managing emotional distress by promoting psychological flexibility. This includes willingness to experience pain-related distress in the pursuit of valued behaviors, engagement in meaningful activities, and improved pain management. ACT can be delivered in brief and modular formats, making it widely applicable, feasible, well tolerated, and effective. As a transdiagnostic approach, ACT targets core processes underlying human suffering, making it potentially suitable for all CPP conditions. Evidence shows that ACT-based treatments effectively reduce pain intensity, pain interference, and emotional distress, while improving patients' quality of life.

However, access to these programs is often limited by healthcare system constraints, shortages of trained professionals, lack of service proximity, stigma associated with psychological treatment, and patients' mobility difficulties. In an effort to enhance the time- and cost-effectiveness of psychological interventions, recent years have seen the development of delivery modes complementing face-to-face treatment. Among these, internet-based self-help interventions grounded in the principles of cognitive-behavioral therapy (CBT) have proven promising for the treatment of chronic pain and related disorders. Using the internet as a delivery format for CBT interventions may potentially overcome many of these barriers.

Some advantages of internet-based interventions (IBIs) include reducing therapist time per patient, shortening waiting lists, enabling patients to work at their own pace, eliminating the need to schedule appointments with a therapist, increasing accessibility to a greater number of patients, and being cost-effective. IBI for chronic pain management has been shown to reduce pain, depression, anxiety, and disability, while improving quality of life. Recently, several studies have implemented IBIs based on ACT principles. Evidence demonstrates that Internet-based Acceptance and Commitment Therapy Interventions can impact pain acceptance, anxiety, depression, catastrophizing, pain interference, affective distress, pain intensity, pain-related disability, and fear-avoidance, with effect sizes ranging from small to large.

Study Objectives

The present study aims to examine the effectiveness, in terms of pain acceptance and cost-effectiveness, of a guided internet-based ACT intervention, implemented and adapted for the Italian population, targeting patients with Chronic Pain. Furthermore, covariates that may moderate or mediate the effects will be investigated in order to gain a deeper understanding of the mechanisms underlying the effects of MobACT. The specific objectives of the study are:

1. To examine the effectiveness of a guided internet-based ACT intervention (MobACT) compared to a waitlist control group, in terms of pain acceptance;
2. To investigate which factors moderate and mediate the effects of a guided internet-based ACT intervention (MobACT);
3. To evaluate the cost-effectiveness of the MobACT intervention.

Method and Analysis

Study Design

A two-group randomized controlled trial will be conducted. Participants will be randomized either to a treatment group or to a waitlist control group, which will receive the treatment after completion of the post-treatment assessments (7 weeks after study initiation). Informed consent will be obtained from all participants.

Measurements Assessments will be collected at three time points using self-administered online questionnaires delivered through the treatment platform: pre-intervention (T0), post-intervention (T1), and 6-month follow-up (T2), the latter only for the experimental group.

Each week, during the seven weeks of the intervention, participants will be presented with a Visual Analogue Scale (VAS) to evaluate their perceived sleep quality during that week ("How would you rate the quality of your sleep during this week?"), ranging from 0 ("the worst imaginable sleep quality") to 100 ("the best imaginable sleep quality"). In addition, participants will be asked to report any changes in their pharmacological therapy for Chronic Pain management on a weekly basis. The item for the first week will read: "Compared to what you reported during the pre-intervention assessment, have there been any changes in your pharmacological therapy for the management of Chronic Pain?" For the subsequent weeks, the item will read: "Compared to the previous week, have there been any changes in your pharmacological therapy for the management of Chronic Pain?"

Response options will be: "No, there have been no changes" and "Yes, there have been changes." If the participant reports changes, they will be asked to specify the type of change: "increased dosage of the same medication(s)," "decreased dosage of the same medication(s)," or "administration of different medication(s)."

Recruitment, Participants, and Randomization

Power Analysis F tests - ANOVA: Repeated measures, within-between interaction Analysis: A priori: Compute required sample size Input: Effect size f = 0.15 α err prob = 0.05 Power (1-β err prob) = 0.95 Number of groups = 2 Number of measurements = 3 Corr among rep measures = 0.5 Nonsphericity correction ε = 1 Output: Noncentrality parameter λ = 15.6600000 Critical F = 3.0354408 Numerator df = 2.0000000 Denominator df = 228 Total sample size = 116 Actual power = 0.9501483

Recruitment

Participants will be recruited online through multiple channels, including social media platforms (e.g., Facebook, Instagram), online support groups, and relevant national and regional patient associations. Online recruitment was chosen to maximize outreach and ensure accessibility for individuals with chronic pain, who may experience mobility limitations and barriers to in-person recruitment. This strategy is expected to enhance the representativeness of the sample by reaching a broad and diverse population, while also ensuring cost-effectiveness and feasibility within the study's timeline and resources.

Inclusion and Exclusion Criteria Since internet-delivered Acceptance and Commitment Therapy (ACT) has proven effective in different groups of patients with Chronic Pain, it has been adapted and implemented according to the study's target population. The inclusion and exclusion criteria for participation are listed below.

Inclusion criteria:

1. Adults aged 18 years or older;
2. A verifiable medical diagnosis of Chronic Pain (duration ≥ 3 months);
3. Internet access;
4. Sufficient competence in the use of computers and the internet;
5. Fluent knowledge of the Italian language.

Exclusion criteria:

1. Current participation in psychological or psychotherapeutic treatments for the management of Chronic Pain;
2. High suicide risk;
3. Cognitive impairments;
4. Presence of clinically certified psychiatric disorders such as:

   1. Psychotic spectrum disorders (schizophrenia, schizoaffective disorders, etc.);
   2. Bipolar disorder (unstabilized manic or hypomanic episodes);
   3. Severe depressive disorders (major depression, suicidal ideation, or recent suicide attempts);
   4. Severe personality disorders, i.e., those preventing the execution of daily activities such as work or self-care;
   5. Cognitive or neurodegenerative disorders.

All participants at high suicide risk, as indicated by a PHQ-9 score ≥ 1 on item nine ("Thoughts that you would be better off dead, or of hurting yourself in some way") and/or a WSQ score ≥ 1 on item fifteen ("Recently, have you had thoughts of harming yourself or taking your own life?"), will be contacted by a therapist. The therapist will provide information about available services and recommend seeking help from their general practitioner, the local Mental Health Center, or an official emergency number.

Online Platform iTerapi The iTerapi platform, developed at Linköping University, is a reliable resource designed to deliver psychological treatments over the internet and conduct research studies, including randomized controlled trials. The platform emphasizes security, process optimization, and personalization, supporting various treatment modalities, including text, audio, and video interactions. Participants access the intervention through a homepage that provides entry to all treatment components using personalized credentials. The platform is designed to be intuitive and user-friendly, ensuring a seamless experience across different devices, including desktops, tablets, and smartphones. The homepage displays new messages and pending questionnaires.

iTerapi ensures data security and confidentiality through encrypted transmission and secure storage of information. Data from each study are isolated, with access restricted to authorized personnel only. Regular backups and system updates are performed to maintain data integrity and platform reliability.

Procedure By accessing the registration link for the MobACT project, participants will first be provided with information about the study, the inclusion and exclusion criteria, the registration process, and instructions on how to access the online modules. After providing informed consent, participants will complete an online screening using specific questionnaires (e.g., WSQ) to confirm their eligibility. Participants will then be invited to a telephone interview with a licensed psychologist-psychotherapist. Following these interviews, the final decision on study participation will be jointly discussed by the clinician and three principal investigators (GC, GP, and MS), based on both quantitative indices and the interview report. The decision regarding inclusion or exclusion will be communicated to participants within a few days.

Eligible participants will be randomized into two groups: an intervention group receiving the MobACT treatment, and a control group (waitlist) that will receive the treatment after seven weeks. A secure online platform, iTerapi, will be used for communication between therapists and participants, program material distribution, and assessment collection. Participants' personal information will be anonymized by assigning each individual a unique code. At the beginning of the intervention, all participants will receive an email containing their username and a personalized link to create their password.

Throughout the program, every Thursday, participants will receive an email notifying them that new material is available. Participants who fail to access the weekly module or complete the exercises will receive a weekly reminder on Monday. This reminder will include a short encouraging message. The treatment program consists of seven modules, delivered weekly, for a total duration of seven weeks. The seven modules cover the following topics:

1. Constructive Despair;
2. Willingness and Pain Acceptance;
3. Defusion from Negative Thoughts;
4. Committed Action and Values;
5. Values and Goals;
6. Willingness Exercises;
7. Maintenance of Learned Strategies.

   At the end of the intervention program, participants in both groups will be asked to complete the post-treatment assessments. Measurements will be conducted at three time points: pre-intervention (T0, baseline), post-intervention (T1, 7-weeks), and 6-month follow-up (T2). During the intervention, participants will also complete weekly assessments of sleep quality and possible changes in pharmacological therapy.

   After the intervention program, approximately 20 participants (until data saturation) assigned to the experimental group will be invited to take part in a brief semi-structured interview, specifically developed to explore their subjective experience with the treatment and technology. Transcriptions of these interviews will undergo qualitative thematic analysis. Data collected will be analyzed using statistical software such as SPSS or R. Analyses will include comparisons between the intervention and control groups in terms of pain acceptance, quality of life, pain intensity, psychological flexibility, and other secondary outcomes.

   Participants will be able to contact a psychologist during the study; however, no scheduled contact will be provided. The system will notify participants that a psychologist will respond to their request within three working days.

   Treatment Program

   The treatment consists of seven modules, each addressing a specific component of Acceptance and Commitment Therapy (ACT). The program follows the procedures recommended by Hayes et al. (1999). The module topics are as follows:

   Constructive Despair: This module introduces the concept of constructive despair. Participants are encouraged to reflect on their efforts to control pain and to acknowledge the ineffectiveness of these attempts. This prepares the ground for acceptance and commitment to new strategies. The "man in the hole" metaphor is used to illustrate these ideas.

   Willingness and Pain Acceptance: Participants learn to distinguish between primary (physical) and secondary (psychological) pain. The concept of willingness and acceptance of pain is introduced. The "shark trap" and "radio" metaphors are used to explain the difference between short-term control and long-term acceptance.

   Defusion from Negative Thoughts: This module focuses on mindfulness and cognitive defusion techniques to help participants separate themselves from negative thoughts and emotions. The "bus" metaphor, where thoughts and emotions are passengers on a bus driven by the participant, is used.

   Committed Action and Values: Participants explore their personal values and learn how to lead a fulfilling life despite pain. The "chessboard" exercise, which distinguishes between the self and psychological content, along with other mindfulness exercises, is used to help participants connect with their values.

   Values and Goals: Building on the previous module, this section helps participants define and commit to actions aligned with their values. Exercises such as the "values compass" and metaphors like "the skier" and "my party" support this process.

   Willingness Exercises: This module provides a variety of exercises to enhance participants' willingness to experience pain without attempting to control it. The "my party" metaphor is used to illustrate mindfulness in daily life and committed action.

   Maintenance of Learned Strategies: The final module involves developing a maintenance plan and reviewing goals established in previous modules. It summarizes the entire program and provides strategies for sustaining the skills learned. Mindfulness practices are emphasized as part of the maintenance plan.

   Measurements and Assessment Tools Participants will complete the Web Screening Questionnaire (WSQ) online during the initial screening phase. The WSQ consists of several items assessing a range of mental health issues, including depression, generalized anxiety disorder (GAD), panic disorder, agoraphobia, specific phobias, social phobia, post-traumatic stress disorder (PTSD), obsessive-compulsive disorder (OCD), alcohol abuse, and suicidal ideation.

   The WSQ is a brief, internet-based instrument comprising 15 items, designed to identify individuals who may have common mental disorders. Developed at the Vrije Universiteit Amsterdam, the WSQ rapidly identifies clinically relevant problems related to mood, anxiety, and alcohol use. The WSQ takes approximately 2 minutes to complete. It will be used in this study to assess participant eligibility according to inclusion and exclusion criteria, ensuring that only participants meeting the requirements proceed to the full evaluation and treatment phases.

   By using the WSQ, the study aims to efficiently and effectively identify participants with common mental disorders, ensuring that those requiring intervention are accurately recognized and directed toward appropriate treatment pathways. The WSQ is ideal for discriminating between individuals with and without a psychiatric condition, as it helps confirm the absence of disorders. However, additional diagnostic procedures are required in cases of positive WSQ screening results.

   Primary Outcome:

   Acceptance of Primary Chronic Pain The Chronic Pain Acceptance Questionnaire (CPAQ) (20 items) is the primary method for quantifying acceptance in populations with Chronic Pain. Each item is rated on a scale from 0 ("Never true") to 6 ("Always true"), where respondents indicate their rating for each item. The CPAQ comprises two subscales: Activity Engagement (AE) and Willingness to Experience Pain (WP). To calculate the CPAQ score, items pertaining to activity engagement and willingness to experience pain are summed to obtain a score for each factor. The total score ranges from 0 to 120 and is obtained by summing the two factor scores. Higher scores indicate higher levels of pain acceptance. The Activity Engagement domain reflects the extent to which patients engage in daily activities regardless of pain, whereas the Willingness to Experience Pain domain reflects the extent to which patients view attempts to avoid or control pain as an ineffective strategy.

   Secondary Outcomes:

   Pain Intensity and Pain Interference

   The Brief Pain Inventory (BPI-I) (10 items) comprises two subscales. The first assesses pain intensity using four Numerical Rating Scales ranging from 0 ("no pain") to 10 ("worst pain imaginable"), evaluating current pain, worst pain, least pain, and average pain over the past 24 hours. The second subscale measures pain interference with general activity, walking, mood, sleep, work, relations with others, and enjoyment of life, using Numerical Rating Scales from 0 ("does not interfere") to 10 ("completely interferes").

   Quality of Life

   The EuroQol-5D-3L (EQ-5D-3L) is a standardized instrument developed to measure quality of life. The questionnaire consists of two parts. The first includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has three severity levels, from 1 ("no problems") to 3 ("extreme problems"). The second part includes a Visual Analogue Scale (EQ VAS) indicating current perceived health status on a scale from 0 ("worst imaginable health") to 100 ("best imaginable health").

   Sleep Quality

   The Mini Sleep Questionnaire (MSQ) (10 items) assesses sleep quality, specifically considering sleep and wakefulness factors. For each item, participants respond on a Numerical Rating Scale from 1 ("Never") to 7 ("Always"), reflecting the option that best describes their past week.

   Central Sensitization The Central Sensitization Inventory (CSI) (35 items) measures current health symptoms related to central sensitization and provides a total score ranging from 0 to 100. Responses range from "never" (0) to "always" (4). Higher scores indicate a greater presence of symptoms associated with central sensitization. A cut-off of 40/100 has shown good sensitivity and specificity for identifying a subgroup of patients with central sensitization syndrome.

   Pain Catastrophizing The Pain Catastrophizing Scale (PCS) (13 items) assesses the level of catastrophic thinking related to pain. Items are rated on a 5-point Likert scale, with 0 indicating "not at all" and 4 indicating "always." The total score ranges from 0 to 52, with higher scores indicating higher levels of pain catastrophizing.

   Psychological Flexibility The Multidimensional Psychological Flexibility Inventory (MPFI-24) is a self-report measure that assesses all flexibility and inflexibility processes within the Hexaflex/Inflexahex model. Using a response scale from 1 ("Never true") to 6 ("Always true"), respondents rate how much each item corresponded to their experience over the past two weeks.

   Self-Efficacy The Pain Self-Efficacy Questionnaire (PSEQ) (10 items) is used in both clinical and research settings to assess pain-related self-efficacy. Patients rate their confidence in performing specific activities despite pain. Each item is rated on a 7-point Likert scale, with 0 indicating "not at all confident" and 6 indicating "completely confident." Total scores are obtained by summing item scores and range from 0 to 60.

   Coping

   The Chronic Pain Coping Inventory (CPCI-42) (42 items) asks patients to rate how often they used behavioral and cognitive coping strategies during the previous week. The Italian version of the CPCI-42, validated across different cultures, confirms its eight-subscale structure. Each subscale yields a score ranging from 0 to 7, with higher scores indicating greater use of the coping strategies.

   Anxiety The Generalized Anxiety Disorder scale (GAD-7) (7 items) includes seven items, each addressing a specific anxiety symptom. Participants indicate how often they were bothered by each symptom over the past 14 days, using a four-point scale: 0 "Not at all," 1 "Several days," 2 "More than half the days," and 3 "Nearly every day." The total score ranges from 0 to 21 (0-4 minimal anxiety, 5-9 mild, 10-14 moderate, 15-21 severe).

   Depression The Patient Health Questionnaire (PHQ-9) is a self-report instrument used to assess depression severity. It comprises nine items, each reflecting a criterion for major depressive disorder as outlined in the DSM-IV. The PHQ-9 asks participants how often they have experienced each symptom over the past two weeks. Items include: little interest or pleasure in doing things; feeling down or hopeless; trouble sleeping or sleeping too much; feeling tired or having little energy; poor appetite or overeating; feeling bad about oneself; trouble concentrating; moving or speaking slowly or being restless; and thoughts of being better off dead or of self-harm. Each item is rated from 0 ("not at all") to 3 ("nearly every day"), with a total score from 0 to 27. Interpretation: 0-4 minimal, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe depression.

   Statistical Analysis The analysis of the primary outcomes aims to evaluate the effectiveness of the MobACT intervention in managing Primary Chronic Pain (PCP). Key outcomes include pain intensity, pain interference, and overall quality of life. The analysis will also examine the intervention's impact on psychological flexibility, emotional distress, and cognitive and behavioral responses to pain.

   Cost-Effectiveness Analysis To conduct the cost-effectiveness analysis, data will be collected from program initiation through the last follow-up, and the resources required to deliver the intervention will be quantified. Patient service utilization will be collected via the MobACT platform, covering the use of additional treatments in hospitals and clinics, other prescribed therapies, hospitalizations, emergency department visits, outpatient visits, service use, medications, and assistive devices.

   To enable an economic evaluation, questionnaires delivered via the iTerapi platform will also collect information on days off work, recreational activities, private expenses (e.g., privately paid therapies, travel costs for care), informal care, benefits received, and lost work hours (including those of family members and friends) related to pain management. The cost-effectiveness analysis will be conducted from both a healthcare sector and a societal perspective, following existing guidelines. The Second Panel on Cost-Effectiveness in Health and Medicine recommends that all studies report a reference analysis from the healthcare sector perspective and another from the societal perspective.

   The Impact Inventory, which lists the health and non-health effects of an intervention, makes the economic evaluation more explicit and transparent. From the healthcare sector perspective, the total program cost per participant will be calculated using a resource costing approach, including personnel, supplies, and equipment costs (e.g., web hosting service, software maintenance) required to deliver MobACT. From the societal perspective, costs will include patient time, transportation, and the cost of lost unpaid productivity due to illness.

   Data Management Data Collection

   Data will be collected using the iTerapi platform, a system designed to deliver psychological treatments and manage research data securely. Participants will access the platform to complete baseline, post-intervention, and follow-up assessments. The platform will be used to administer self-report questionnaires and collect response data in real time.

   Data Storage

   Secure Storage: All data collected via the iTerapi platform will be stored on secure servers with encrypted transmission to protect against unauthorized access. The platform uses industry-standard encryption methods to ensure data security.

   Access Control: Data access will be restricted to authorized study personnel only. Each user will have unique login credentials, and access levels will be assigned based on their study role. This ensures that only those with a legitimate need can view or modify data.

   Data Handling

   Data Entry and Verification: Data entry will be automated through the iTerapi platform, minimizing the risk of manual entry errors.

   Data Confidentiality

   Confidentiality: All participant data will be de-identified prior to analysis. Personally identifiable information, such as email addresses and phone numbers, will be stored separately from research data and linked via a unique participant ID.

   Confidentiality Agreements: All study personnel will be required to sign confidentiality agreements to ensure they understand and commit to protecting participant privacy.

   Data Sharing and Publication: Data will be shared and reported only in aggregate form, without personally identifiable information in any publication or presentation.

   Data Analysis Plan

   Statistical Methods: Statistical analyses will be conducted using appropriate methods to compare outcomes between the intervention and control groups at each assessment point (T0, T1, T2).

   Software: Data analysis will be performed using statistical software such as SPSS, Jamovi, or R, to ensure accuracy and reliability of results.

   Data Cleaning: Prior to analysis, data will be cleaned to remove incomplete or inconsistent entries. This process will include checking for outliers and appropriately handling missing data.

   Data Access and Retention

   Access Protocol: Data access will be strictly controlled and documented. Only authorized personnel involved in the analysis and oversight of the study will have access.

   Retention Period: Data will be retained for a period specified by institutional policies and regulatory requirements, typically for at least five years after study completion. After this period, data will be archived or securely destroyed in accordance with policies.

   Expected Results

   Over the past decade, internet-based cognitive behavioral therapy (ICBT) has been developed and tested in numerous controlled studies, and more recently several studies have implemented internet-delivered interventions grounded in ACT principles. Owing to its characteristics, this therapeutic approach may be useful in supporting patients with Chronic Pain: Hughes et al. (2017) and Veehof et al. (2016) emphasize that ACT-based treatments effectively reduce pain intensity, pain interference, and emotional distress, thereby improving patients' quality of life. This intervention is expected to be feasible and effective in improving acceptance of Chronic Pain, quality of life and sleep, psychological flexibility, self-efficacy, coping, and the management of anxiety and/or depressive symptoms, as well as in reducing pain intensity and interference, the heightened responsiveness of the central nervous system to stimuli, and the level of catastrophic thoughts associated with pain.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older;
2. A verifiable medical diagnosis of Chronic Pain (duration ≥ 3 months);
3. Internet access;
4. Sufficient computer and internet literacy;
5. Fluent knowledge of the Italian language.

Exclusion Criteria:

1. Current participation in psychological or psychotherapeutic treatments for chronic pain management;
2. High risk of suicide;
3. Cognitive impairments;
4. Presence of certified psychiatric disorders, such as:

   1. Psychotic disorders (e.g., schizophrenia, schizoaffective disorders, etc.);
   2. Bipolar disorder (unstabilized manic or hypomanic episodes);
   3. Severe depressive disorders (e.g., major depression, suicidal intent, or recent suicide attempts);
   4. Severe personality disorders that impair the ability to carry out daily activities (e.g., work, self-care);
   5. Cognitive or neurodegenerative disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Acceptance of Chronic Pain | T0 (baseline); T1 (7-weeks); T2 (6 months)
  The Chronic Pain Acceptance Questionnaire (CPAQ) (20 items) is the primary method used to assess acceptance in individuals with chronic pain. Each item is rated on a scale from 0 ("Never true") to 6 ("Always true"), where the respondent indicates their level of agreement with each statement.
  The CPAQ is composed of two subscales: Activity Engagement (AE) and Pain Willingness (PW). To calculate the CPAQ score, the items corresponding to each subscale are summed to obtain a score for each domain. The total score, ranging from 0 to 120, is the sum of the two subscale scores. Higher scores indicate greater levels of pain acceptance.
  The Activity Engagement (AE) subscale measures the extent to which individuals continue to engage in daily activities regardless of their pain, while the Pain Willingness (PW) subscale assesses the extent to which individuals perceive that avoiding or controlling pain is an ineffective strategy.

SECONDARY OUTCOMES:
Pain Intensity and Pain Interference | T0 (baseline); T1 (7-weeks); T2 (6 months)
  The Brief Pain Inventory - Italian version (BPI-I) (10 items) consists of two subscales.
  The first subscale assesses pain intensity using four Numerical Rating Scales, ranging from 0 ("no pain") to 10 ("pain as bad as you can imagine"), which measure current pain, worst pain, least pain, and average pain experienced over the past 24 hours.
  The second subscale evaluates pain interference with various aspects of daily life, including general activity, walking, mood, sleep, work, relationships with others, and enjoyment of life. These are also rated on Numerical Rating Scales from 0 ("does not interfere") to 10 ("completely interferes").
  The Italian version of the BPI has shown good internal consistency (Cronbach's alpha = 0.80), stability (rho = 0.789, p < 0.001), excellent inter-rater reliability (k = 0.945), and good homogeneity (alpha = 0.8).
Quality of Life | T0 (baseline); T1 (7-weeks); T2 (6 months)
  The EuroQol-5D-3L (EQ-5D-3L) is a standardized instrument developed to assess quality of life. The questionnaire consists of two parts. The first part includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each rated on three levels of severity, from 1 ("no problems") to 3 ("extreme problems"). The second part features a Visual Analogue Scale (EQ VAS) that assesses the respondent's current perceived health on a scale from 0 ("worst imaginable health") to 100 ("best imaginable health").
  The Italian version of the EQ-5D-3L has shown good reliability, with a Cronbach's alpha coefficient of 0.73.
Sleep Quality | T0 (baseline); T1 (7-weeks); T2 (6 months)
  The Mini Sleep Questionnaire (MSQ) (10 items) evaluates sleep quality by assessing both sleep and wakefulness factors. Each item is rated on a Numerical Rating Scale (NRS) from 1 ("Never") to 7 ("Always"), referring to the respondent's experience over the past week.
  The Italian version of the MSQ has demonstrated good internal consistency (Cronbach's alpha = 0.77), good test-retest reliability (ICC = 0.82), and factor analysis confirmed two dimensions (sleep and wakefulness) with Cronbach's alpha = 0.75 for both. Optimal cut-off values were identified (>16 for sleep and >14 for wakefulness), with an area under the curve greater than 0.80.
Central Sensitization | T0 (baseline); T1 (7-weeks); T2 (6 months)
  The Central Sensitization Inventory (CSI) (35 items) measures current health symptoms related to central sensitization, yielding a total score ranging from 0 to 100. Items are rated on a scale from "never" (0) to "always" (4), with higher scores indicating greater presence of central sensitization symptoms. A cut-off score of 40 has demonstrated good sensitivity and specificity for identifying patients with central sensitization syndromes.
  The Italian version of the CSI has shown good internal consistency (Cronbach's alpha = 0.87), ranging from 0.86 to 0.87 when individual items are removed.
Pain Catastrophizing | T0 (baseline); T1 (7-weeks); T2 (6 months)
  The Pain Catastrophizing Scale (PCS) (13 items) is used to assess the level of catastrophizing thoughts associated with pain. Each item is rated on a 5-point Likert scale, from 0 ("not at all") to 4 ("all the time"). The total score ranges from 0 to 52, with higher scores indicating greater pain catastrophizing.
  The Italian version of the PCS has demonstrated excellent internal consistency (Cronbach's alpha = 0.92) and test-retest reliability (ICC = 0.842, p < 0.001).
Psychological Flexibility | T0 (baseline); T1 (7-weeks); T2 (6 months)
  The Multidimensional Psychological Flexibility Inventory (MPFI-24) is a self-report measure assessing all flexibility and inflexibility processes within the Hexaflex/Inflexahex model. Respondents rate how well each item reflects their experience over the past two weeks using a 6-point Likert scale from 1 ("Never true") to 6 ("Always true").
  The Italian version of the MPFI has demonstrated excellent internal consistency (Cronbach's alpha = 0.94) for both overall psychological flexibility and inflexibility, with subscale alphas ranging from 0.85 to 0.94.
Self-Efficacy | T0 (baseline); T1 (7-weeks); T2 (6 months)
  The Pain Self-Efficacy Questionnaire (PSEQ) (10 items) is used in both clinical and research contexts to assess individuals' confidence in performing activities despite pain. Each item is rated on a 7-point Likert scale, from 0 ("not at all confident") to 6 ("completely confident"). Total scores range from 0 to 60, with higher scores indicating greater pain-related self-efficacy.
  The Italian version of the PSEQ has shown excellent internal consistency (Cronbach's alpha = 0.94) and good test-retest reliability (ICC = 0.82).
Coping | T0 (baseline); T1 (7-weeks); T2 (6 months)
  The Chronic Pain Coping Inventory (CPCI-42) (42 items) asks patients to rate how often they used behavioral and cognitive coping strategies during the previous week. The Italian version, validated across cultures, maintains its eight-subscale structure, with each subscale producing a score from 0 to 7. Higher scores reflect more frequent use of coping strategies.
  The Italian CPCI-42 has shown good internal consistency (Cronbach's alpha = 0.71-0.80) and reliability (ICC = 0.70-0.85, and >0.85 for all subscales).
Anxiety | T0 (baseline); T1 (7-weeks); T2 (6 months)
  The Generalized Anxiety Disorder scale (GAD-7) (7 items) assesses symptoms of generalized anxiety. Respondents rate how often they have been bothered by each symptom over the past 14 days on a 4-point scale: 0 ("Not at all"), 1 ("Several days"), 2 ("More than half the days"), and 3 ("Nearly every day"). Total scores range from 0 to 21 and are interpreted as follows: 0-4 = minimal anxiety, 5-9 = mild anxiety, 10-14 = moderate anxiety, 15-21 = severe anxiety.
  The Italian version of the GAD-7 has shown good internal consistency (Cronbach's alpha = 0.918) and test-retest reliability (ICC = 0.83).
Depression | T0 (baseline); T1 (7-weeks); T2 (6 months)
  The Patient Health Questionnaire (PHQ-9) is a self-report measure used to assess the severity of depressive symptoms. The nine items correspond to the DSM-IV criteria for major depressive disorder and evaluate symptom frequency over the past two weeks. Items include: little interest or pleasure in doing things, feeling down or hopeless, sleep issues, fatigue, appetite changes, feelings of worthlessness, difficulty concentrating, psychomotor changes, and suicidal thoughts. Each item is scored from 0 ("Not at all") to 3 ("Nearly every day"), with total scores ranging from 0 to 27. Interpretation: 0-4 = minimal depression, 5-9 = mild, 10-14 = moderate, 15-19 = moderately severe, and 20-27 = severe depression.
  The Italian version of the PHQ-9 has demonstrated good internal consistency (Cronbach's alpha = 0.918).

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Castelnuovo, Ph.D., Principal Investigator — Catholic University of Sacred Heart of Milan
Locations (4):
- Italy (3):
  - Alma Mater Studiorum of Bologna, Bologna
  - Catholic University of Sacred Heart, Milan
  - University of Verona, Verona
- University of Linkoping, Linköping, Sweden

REFERENCES:
- [Background] Vugts MAP, Joosen MCW, van der Geer JE, Zedlitz AMEE, Vrijhoef HJM. The effectiveness of various computer-based interventions for patients with chronic pain or functional somatic syndromes: A systematic review and meta-analysis. PLoS One. 2018 May 16;13(5):e0196467. doi: 10.1371/journal.pone.0196467. eCollection 2018. PMID 29768436
- [Background] Vlaescu G, Alasjo A, Miloff A, Carlbring P, Andersson G. Features and functionality of the Iterapi platform for internet-based psychological treatment. Internet Interv. 2016 Oct 3;6:107-114. doi: 10.1016/j.invent.2016.09.006. eCollection 2016 Nov. PMID 30135819
- [Background] Sleed M, Eccleston C, Beecham J, Knapp M, Jordan A. The economic impact of chronic pain in adolescence: methodological considerations and a preliminary costs-of-illness study. Pain. 2005 Dec 15;119(1-3):183-190. doi: 10.1016/j.pain.2005.09.028. Epub 2005 Nov 16. PMID 16297552
- [Background] Scott W, Hann KE, McCracken LM. A Comprehensive Examination of Changes in Psychological Flexibility Following Acceptance and Commitment Therapy for Chronic Pain. J Contemp Psychother. 2016;46:139-148. doi: 10.1007/s10879-016-9328-5. Epub 2016 Mar 2. PMID 27397934
- [Background] Schutze R, Rees C, Smith A, Slater H, Campbell JM, O'Sullivan P. How Can We Best Reduce Pain Catastrophizing in Adults With Chronic Noncancer Pain? A Systematic Review and Meta-Analysis. J Pain. 2018 Mar;19(3):233-256. doi: 10.1016/j.jpain.2017.09.010. Epub 2017 Nov 6. PMID 29122652
- [Background] Savoia E, Fantini MP, Pandolfi PP, Dallolio L, Collina N. Assessing the construct validity of the Italian version of the EQ-5D: preliminary results from a cross-sectional study in North Italy. Health Qual Life Outcomes. 2006 Aug 10;4:47. doi: 10.1186/1477-7525-4-47. PMID 16901340
- [Background] Sanders GD, Neumann PJ, Basu A, Brock DW, Feeny D, Krahn M, Kuntz KM, Meltzer DO, Owens DK, Prosser LA, Salomon JA, Sculpher MJ, Trikalinos TA, Russell LB, Siegel JE, Ganiats TG. Recommendations for Conduct, Methodological Practices, and Reporting of Cost-effectiveness Analyses: Second Panel on Cost-Effectiveness in Health and Medicine. JAMA. 2016 Sep 13;316(10):1093-103. doi: 10.1001/jama.2016.12195. PMID 27623463
- [Background] Pietrabissa G, Semonella M, Marchesi G, Mannarini S, Castelnuovo G, Andersson G, Rossi AA. Validation of the Italian Version of the Web Screening Questionnaire for Common Mental Disorders. J Clin Med. 2024 Feb 19;13(4):1170. doi: 10.3390/jcm13041170. PMID 38398481
- [Background] Perlini C, Donisi V, Rossetti MG, Moltrasio C, Bellani M, Brambilla P. The potential role of EMDR on trauma in affective disorders: A narrative review. J Affect Disord. 2020 May 15;269:1-11. doi: 10.1016/j.jad.2020.03.001. Epub 2020 Mar 14. PMID 32217337
- [Background] Pakenham KI, Landi G, Boccolini G, Furlani A, Grandi S, Tossani E. The moderating roles of psychological flexibility and inflexibility on the mental health impacts of COVID-19 pandemic and lockdown in Italy. J Contextual Behav Sci. 2020 Jul;17:109-118. doi: 10.1016/j.jcbs.2020.07.003. Epub 2020 Jul 20. PMID 32834969
- [Background] Nicholas M, Vlaeyen JWS, Rief W, Barke A, Aziz Q, Benoliel R, Cohen M, Evers S, Giamberardino MA, Goebel A, Korwisi B, Perrot S, Svensson P, Wang SJ, Treede RD; IASP Taskforce for the Classification of Chronic Pain. The IASP classification of chronic pain for ICD-11: chronic primary pain. Pain. 2019 Jan;160(1):28-37. doi: 10.1097/j.pain.0000000000001390. PMID 30586068
- [Background] Monticone M, Ferrante S, Rocca B, Nava T, Parini C, Cerri C. Chronic pain acceptance questionnaire: confirmatory factor analysis, reliability, and validity in Italian subjects with chronic low back pain. Spine (Phila Pa 1976). 2013 Jun 1;38(13):E824-31. doi: 10.1097/BRS.0b013e3182917299. PMID 23524871
- [Background] Monticone M, Baiardi P, Ferrari S, Foti C, Mugnai R, Pillastrini P, Rocca B, Vanti C. Development of the Italian version of the Pain Catastrophising Scale (PCS-I): cross-cultural adaptation, factor analysis, reliability, validity and sensitivity to change. Qual Life Res. 2012 Aug;21(6):1045-50. doi: 10.1007/s11136-011-0007-4. Epub 2011 Sep 13. PMID 21912846
- [Background] Macea DD, Gajos K, Daglia Calil YA, Fregni F. The efficacy of Web-based cognitive behavioral interventions for chronic pain: a systematic review and meta-analysis. J Pain. 2010 Oct;11(10):917-29. doi: 10.1016/j.jpain.2010.06.005. Epub 2010 Jul 22. PMID 20650691
- [Background] Lin J, Paganini S, Sander L, Luking M, Ebert DD, Buhrman M, Andersson G, Baumeister H. An Internet-Based Intervention for Chronic Pain. Dtsch Arztebl Int. 2017 Oct 13;114(41):681-688. doi: 10.3238/arztebl.2017.0681. PMID 29082858
- [Background] Landi G, Furlani A, Boccolini G, Mikulincer M, Grandi S, Tossani E. Tolerance for Mental Pain Scale (TMPS): Italian validation and evaluation of its protective role in depression and suicidal ideation. Psychiatry Res. 2020 Sep;291:113263. doi: 10.1016/j.psychres.2020.113263. Epub 2020 Jun 30. PMID 32623264
- [Background] Hughes LS, Clark J, Colclough JA, Dale E, McMillan D. Acceptance and Commitment Therapy (ACT) for Chronic Pain: A Systematic Review and Meta-Analyses. Clin J Pain. 2017 Jun;33(6):552-568. doi: 10.1097/AJP.0000000000000425. PMID 27479642
- [Background] Heapy AA, Higgins DM, Cervone D, Wandner L, Fenton BT, Kerns RD. A Systematic Review of Technology-assisted Self-Management Interventions for Chronic Pain: Looking Across Treatment Modalities. Clin J Pain. 2015 Jun;31(6):470-92. doi: 10.1097/AJP.0000000000000185. PMID 25411862
- [Background] Hayes SC, Wilson KG, Gifford EV, Follette VM, Strosahl K. Experimental avoidance and behavioral disorders: a functional dimensional approach to diagnosis and treatment. J Consult Clin Psychol. 1996 Dec;64(6):1152-68. doi: 10.1037//0022-006x.64.6.1152. PMID 8991302
- [Background] Golfieri L, Gitto S, Vukotic R, Andreone P, Marra F, Morelli MC, Cescon M, Grandi S. Impact of psychosocial status on liver transplant process. Ann Hepatol. 2019 Nov-Dec;18(6):804-809. doi: 10.1016/j.aohep.2019.06.011. Epub 2019 Aug 20. PMID 31471202
- [Background] Giusti EM, Pietrabissa G, Manzoni GM, Cattivelli R, Molinari E, Trompetter HR, Schreurs KMG, Castelnuovo G. The Economic Utility of Clinical Psychology in the Multidisciplinary Management of Pain. Front Psychol. 2017 Oct 31;8:1860. doi: 10.3389/fpsyg.2017.01860. eCollection 2017. No abstract available. PMID 29163260
- [Background] Gasslander N, Andersson G, Bostrom F, Brandelius L, Pelling L, Hamrin L, Gordh T, Buhrman M. Tailored internet-based cognitive behavioral therapy for individuals with chronic pain and comorbid psychological distress: a randomized controlled trial. Cogn Behav Ther. 2022 Sep;51(5):408-434. doi: 10.1080/16506073.2022.2065528. Epub 2022 May 9. PMID 35533363
- [Background] Gandy M, Pang STY, Scott AJ, Heriseanu AI, Bisby MA, Dudeney J, Karin E, Titov N, Dear BF. Internet-delivered cognitive and behavioural based interventions for adults with chronic pain: a systematic review and meta-analysis of randomized controlled trials. Pain. 2022 Oct 1;163(10):e1041-e1053. doi: 10.1097/j.pain.0000000000002606. Epub 2022 Feb 7. PMID 35121696
- [Background] Gallego A, Serrat M, Royuela-Colomer E, Sanabria-Mazo JP, Borras X, Esteve M, Grasa M, Rosa A, Rozadilla-Sacanell A, Almirall M, D'Amico F, Dai Y, Rosenbluth MJ, McCracken LM, Navarrete J, Feliu-Soler A, Luciano JV. Study protocol for a three-arm randomized controlled trial investigating the effectiveness, cost-utility, and physiological effects of a fully self-guided digital Acceptance and Commitment Therapy for Spanish patients with fibromyalgia. Digit Health. 2024 Mar 27;10:20552076241239177. doi: 10.1177/20552076241239177. eCollection 2024 Jan-Dec. PMID 38550263
- [Background] Feliu-Soler A, Montesinos F, Gutierrez-Martinez O, Scott W, McCracken LM, Luciano JV. Current status of acceptance and commitment therapy for chronic pain: a narrative review. J Pain Res. 2018 Oct 2;11:2145-2159. doi: 10.2147/JPR.S144631. eCollection 2018. PMID 30323649
- [Background] Eccleston C, Fisher E, Craig L, Duggan GB, Rosser BA, Keogh E. Psychological therapies (Internet-delivered) for the management of chronic pain in adults. Cochrane Database Syst Rev. 2014 Feb 26;2014(2):CD010152. doi: 10.1002/14651858.CD010152.pub2. PMID 24574082
- [Background] Chiarotto A, Viti C, Sulli A, Cutolo M, Testa M, Piscitelli D. Cross-cultural adaptation and validity of the Italian version of the Central Sensitization Inventory. Musculoskelet Sci Pract. 2018 Oct;37:20-28. doi: 10.1016/j.msksp.2018.06.005. Epub 2018 Jun 15. PMID 29966856
- [Background] Chiarotto A, Vanti C, Ostelo RW, Ferrari S, Tedesco G, Rocca B, Pillastrini P, Monticone M. The Pain Self-Efficacy Questionnaire: Cross-Cultural Adaptation into Italian and Assessment of Its Measurement Properties. Pain Pract. 2015 Nov;15(8):738-47. doi: 10.1111/papr.12242. Epub 2014 Sep 27. PMID 25264358
- [Background] Cattivelli R, Castelnuovo G, Musetti A, Varallo G, Spatola CAM, Riboni FV, Usubini AG, Tosolin F, Manzoni GM, Capodaglio P, Rossi A, Pietrabissa G, Molinari E. ACTonHEALTH study protocol: promoting psychological flexibility with activity tracker and mHealth tools to foster healthful lifestyle for obesity and other chronic health conditions. Trials. 2018 Nov 29;19(1):659. doi: 10.1186/s13063-018-2968-x. PMID 30486868
- [Background] Caraceni A, Mendoza TR, Mencaglia E, Baratella C, Edwards K, Forjaz MJ, Martini C, Serlin RC, de Conno F, Cleeland CS. A validation study of an Italian version of the Brief Pain Inventory (Breve Questionario per la Valutazione del Dolore). Pain. 1996 Apr;65(1):87-92. doi: 10.1016/0304-3959(95)00156-5. PMID 8826494
- [Background] Buhrman M, Skoglund A, Husell J, Bergstrom K, Gordh T, Hursti T, Bendelin N, Furmark T, Andersson G. Guided internet-delivered acceptance and commitment therapy for chronic pain patients: a randomized controlled trial. Behav Res Ther. 2013 Jun;51(6):307-15. doi: 10.1016/j.brat.2013.02.010. Epub 2013 Mar 14. PMID 23548250
- [Background] Bendelin N, Bjorkdahl P, Risell M, Nelson KZ, Gerdle B, Andersson G, Buhrman M. Patients' experiences of internet-based Acceptance and commitment therapy for chronic pain: a qualitative study. BMC Musculoskelet Disord. 2020 Apr 6;21(1):212. doi: 10.1186/s12891-020-03198-1. PMID 32252707
- [Background] Ariza-Mateos, M. J., Cabrera-Martos, I., Prados-Román, E., Granados-Santiago, M., Rodríguez-Torres, J., & Valenza, M. C. (2021). A systematic review of internet-based interventions for women with chronic pain. British Journal of Occupational Therapy, 84(1),6-14. doi:10.1177/0308022620970861